CLINICAL TRIAL: NCT01718145
Title: A Phase 3, Comparative Study of Asunaprevir and Daclatasvir (DUAL) Combination Therapy Versus Telaprevir Therapy in Japanese Genotype 1b Chronic Hepatitis C IFN Eligible-naive Subjects With a Single Arm Assessment of DUAL Therapy in IFN-therapy Relapsers
Brief Title: A Phase 3, Comparative Study of Asunaprevir and Daclatasvir Combination Therapy Versus Telaprevir Therapy in Japanese HCV Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI447-031
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; asunaprevir; Ribavirin; telaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: Daclatasvir + Asunaprevir (Experimental): Daclatasvir 60 mg tablets by mouth once daily and Asunaprevir 200 mg capsules by mouth twice daily for 24 weeks
  - Naive cohort
  Interventions: Drug: Daclatasvir; Drug: Asunaprevir
- Arm 2: Telaprevir + pegIFNα-2b + Ribavirin (Active Comparator): Telaprevir 750 mg tablets by mouth three times daily, pegIFNα-2b 1.5 μg/kg solution by Subcutaneous weekly & Ribavirin 600- 1000 mg Capsules by mouth twice daily for 24 Weeks
  - Naive cohort
  Interventions: Drug: Ribavirin; Biological: pegIFNα-2b; Drug: Telaprevir
- Arm 3: Daclatasvir + Asunaprevir (Experimental): Daclatasvir 60 mg tablets by mouth once daily and Asunaprevir 200 mg capsules by mouth twice daily for 24 weeks
  - Relapser cohort
  Interventions: Drug: Daclatasvir; Drug: Asunaprevir

INTERVENTIONS:
Drug: Daclatasvir
  Arms: Arm 1: Daclatasvir + Asunaprevir; Arm 3: Daclatasvir + Asunaprevir
Drug: Asunaprevir
  Arms: Arm 1: Daclatasvir + Asunaprevir; Arm 3: Daclatasvir + Asunaprevir
Drug: Ribavirin
  Arms: Arm 2: Telaprevir + pegIFNα-2b + Ribavirin
Biological: pegIFNα-2b
  Arms: Arm 2: Telaprevir + pegIFNα-2b + Ribavirin
Drug: Telaprevir
  Arms: Arm 2: Telaprevir + pegIFNα-2b + Ribavirin

SUMMARY:
The purpose of this study is to assess the anti-viral activity of BMS-790052 and BMS-650032 combination therapy in Japanese subject.

The purpose of this study is to compare the anti-viral activity of the co-administration of Asunaprevir (ASV) and Daclatasvir (DCV) to Telaprevir (TVR) included therapy in Japanese Hepatitis C virus (HCV) subjects

DETAILED DESCRIPTION:
Intervention Model: Parallel in the Naive cohort and Single group in the Relapser cohort

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV-1b infected patient
* HCV Ribonucleic acid (RNA) > 100,000 IU/mL at screening
* Ages 20 to 70 years (for the Naive cohort), ages 20 to 75 years (for the Relapser cohort)
* Treatment naive subjects to Interferon (IFN) based therapy
* Subjects who had undetectable HCV RNA at end of treatment with prior exposure to an IFN-containing regimen, but HCV RNA detectable within 24 weeks of treatment follow-up

Exclusion Criteria:

* Patients who have;

  * Hepatocellular carcinoma
  * Co-infection with Hepatitis B virus (HBV) or Human immunodeficiency virus (HIV)
  * Severe or uncontrollable complication

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with SVR12, defined as HCV RNA target detected or target not detected below LLOQ in the naive cohort | After 12 weeks of the last dose
  * SVR12 = Sustained virologic response at post-treatment Week 12
  * LLOQ = Lower Limit of quantitation

SECONDARY OUTCOMES:
Proportion of subjects with hemoglobin < 10g/dL | First 12 weeks of treatment
Proportion of subjects with rash-related dermatologic events | First 12 weeks of treatment
Proportion of subjects with HCV RNA target detected or target not detected below LLOQ in the naive cohort | At weeks 1, 2, 4, 6, 8 and 12; at both Weeks 4 and 12; EOT (up to 24 weeks), post-treatment Week 4 and post-treatment Week 24
  EOT = End of treatment
Proportion of subjects with HCV RNA target not detected in the naive cohort | At weeks 1, 2, 4, 6, 8 and 12; at both Weeks 4 and 12 [eRVR]; EOT (up to 24 weeks), post-treatment Week 4, post-treatment Week 12 and post-treatment Week 24
  eRVR = Extended rapid virologic response
Proportion of subjects with SVR12, defined as HCV RNA target detected or target not detected below LLOQ in the relapser cohort | At post-treatment Week 12
Proportion of subjects with HCV RNA target detected or target not detected below LLOQ in the relapser cohort | At weeks 1, 2, 4, 6, 8 and 12; at both Weeks 4 and 12; EOT (up to 24 weeks), post-treatment Week 4 and Week 24
Proportion of subjects with HCV RNA target not detected in the relapser cohort | At weeks 1, 2, 4, 6, 8 and 12; at both Weeks 4 and 12 [eRVR]; EOT (up to 24 weeks), post-treatment Week 4, post-treatment Week 12 and post-treatment Week 24
On treatment safety, as measured by the frequency of Severe adverse events (SAEs), discontinuation and dose modification/interruption due to Adverse events (AEs), Grade 3-4 abnormalities observed from clinical laboratory tests for each treatment group | End of treatment (24 weeks) plus 7days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (41):
- Japan (41):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Toyoake Shi, Aichi-ken
  - Local Institution, Chiba, Chiba
  - Local Institution, Fukui-shi, Fukui
  - Local Institution, Fukuoka, Fukuoka
  - Local Institution, Kurume, Fukuoka
  - Local Institution, Gifu, Gifu
  - Local Institution, Ogaki-shi, Gifu
  - Local Institution, Takasaki, Gunma
  - Local Institution, Hiroshima, Hiroshima
  - Local Institution, Obihiro-shi, Hokkaido
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Takamatsu, Kagawa-ken
  - Local Institution, Kagoshima, Kagoshima-ken
  - Local Institution, Kawasaki-shi, Kanagawa
  - Local Institution, Yokohama, Kanagawa
  - Local Institution, Kumamoto, Kumamoto
  - Local Institution, Kyoto, Kyoto
  - Local Institution, Sendai, Miyagi
  - Local Institution, Matsumoto, Nagano
  - Local Institution, Nagasaki, Nagasaki
  - Local Institution, Ōmura, Nagasaki
  - Local Institution, Kashihara, Nara
  - Local Institution, Yufu, Oita Prefecture
  - Local Institution, Okayama, Okayama-ken
  - Local Institution, Osaka, Osaka
  - Local Institution, Osaka-sayama-shi, Osaka
  - Local Institution, Suita, Osaka
  - Local Institution, Suita-shi, Osaka
  - Local Institution, Iruma-gun, Saitama
  - Local Institution, Saitama, Saitama
  - Local Institution, Izunokuni, Shizuoka
  - Local Institution, Shimotsuke-shi, Tochigi
  - Local Institution, Bunkyo-ku, Tokyo
  - Local Institution, Minato-ku, Tokyo
  - Local Institution, Musashino-shi, Tokyo
  - Local Institution, Shinagawa-ku, Tokyo
  - Local Institution, Yamagata, Yamagata
  - Local Institution, Chuo-shi, Yamanashi
  - Local Institution, Nagoya
  - Local Institution, Nishinomiya-shi

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx